CLINICAL TRIAL: NCT01626443
Title: Role of Myo-inositol and D-chiro Inositol on the Ovaric and Metabolic Functions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MI-DCI
Record Dates: First submitted 2012-06-15; First posted 2012-06-22 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: PCOS
Keywords: PCOS; Metabolic disorders; Ovarian functionality; Myo-inositol; D-chiro-inositol
MeSH Terms: conditions — Metabolic Diseases | interventions — Inositol; Folic Acid

ARMS (2):
- Folic acid (Active Comparator)
  Interventions: Dietary Supplement: Folic acid
- Inofolic Combi (Experimental)
  Interventions: Dietary Supplement: Myo-inositol + D-chiro-inositol + Folic acid

INTERVENTIONS:
Dietary Supplement: Myo-inositol + D-chiro-inositol + Folic acid — Myo-inositol (550 mg) + D-chiro-inositol (13.8 mg) + Folic acid (200 mcg); 2 x die
  Arms: Inofolic Combi
Dietary Supplement: Folic acid — Folic acid (200 mcg); 2 x die
  Arms: Folic acid

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine disorders in women of reproductive age and is characterized by menstrual abnormalities, clinical or biochemical hyperandrogenism, multiple abnormal cysts and enlarge ovaries. Women affected by PCOS often suffer of insulin resistance and of a compensatory hyperinsulinemia which put them at risk of developing several metabolic disorders. Inositol is a six-carbon polyol which has been characterized as an insulin sensitizer: it exists as nine different isomers and among them myo-inositol and D-chiroinositol are the most represented and studied in physiology and physiopathology. In particular, myo-inositol (MI) and D-chiro inositol (DCI) glycans administration has been reported to exert beneficial effects at metabolic, hormonal and ovarian levels.

The aim of this randomized study is to evaluate the metabolic and ovaric effects of a six-month supplementation of myo-inositol and D-chiro-inositol on young women with PCOS and hyperinsulemia.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Women aged between 14-40 years
* BMI > 28
* Hyperinsulinemia

Exclusion Criteria:

* Pre-existing secondary endocrine and metabolic disorders
* Pre-existing secondary adrenal disorders
* Pharmacologic treatment in the last 3 months before entering the study
* Pregnancy

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Menstrual cycle restoration | At 6 months
Score hirsutism (Ferriman-Gallwey classification) | At 6 months
Serum progesterone | At 6 months
Testosterone level test | At 6 months
Oral glucose tolerance test (OGTT) | At 6 months
  Evaluation of glycemia and insulinemia levels
Homeostasis Model Assessment (HOMA-index) | At 6 months
Sex hormone binding globulin (SHBG) test | At 6 months
Androstenediol level test | At 6 months
Androstenedione level test | At 6 months
Free Androgen Index (FAI) level test | At 6 months

SECONDARY OUTCOMES:
Body Mass Index (BMI) | At 6 months
Change from baseline in diastolic blood pressure levels | At 6 months
Change from baseline in systolic blood pressure levels | At 6 months
Number of patients with abnormal ovarian size and morphology | At 6 months
  Ovarian ultrasound scan for the assessment of size and morphology
Luteinizing Hormone (LH) level test | At 6 months
  Analysis of LH levels should be performed between the 7th and the 10th day of the cycle
Follicle Stimulating Hormone (FSH) level test | At 6 months
  Analysis of FSH levels should be performed between the 7th and the 10th day of the cycle
Estradiol (E2) level test | At 6 months
  Analysis of E2 levels should be performed between the 7th and the 10th day of the cycle

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa - Department of Endocrinology, Pisa, Italy

REFERENCES:
- [Background] Diamanti-Kandarakis E, Kouli CR, Bergiele AT, Filandra FA, Tsianateli TC, Spina GG, Zapanti ED, Bartzis MI. A survey of the polycystic ovary syndrome in the Greek island of Lesbos: hormonal and metabolic profile. J Clin Endocrinol Metab. 1999 Nov;84(11):4006-11. doi: 10.1210/jcem.84.11.6148. PMID 10566641
- [Background] Nestler JE. Role of hyperinsulinemia in the pathogenesis of the polycystic ovary syndrome, and its clinical implications. Semin Reprod Endocrinol. 1997 May;15(2):111-22. doi: 10.1055/s-2007-1016294. PMID 9165656
- [Background] Baillargeon JP, Nestler JE, Ostlund RE, Apridonidze T, Diamanti-Kandarakis E. Greek hyperinsulinemic women, with or without polycystic ovary syndrome, display altered inositols metabolism. Hum Reprod. 2008 Jun;23(6):1439-46. doi: 10.1093/humrep/den097. Epub 2008 Mar 29. PMID 18375940
- [Background] Nestler JE, Jakubowicz DJ, Reamer P, Gunn RD, Allan G. Ovulatory and metabolic effects of D-chiro-inositol in the polycystic ovary syndrome. N Engl J Med. 1999 Apr 29;340(17):1314-20. doi: 10.1056/NEJM199904293401703. PMID 10219066
- [Background] Chiu TT, Rogers MS, Law EL, Briton-Jones CM, Cheung LP, Haines CJ. Follicular fluid and serum concentrations of myo-inositol in patients undergoing IVF: relationship with oocyte quality. Hum Reprod. 2002 Jun;17(6):1591-6. doi: 10.1093/humrep/17.6.1591. PMID 12042283
- [Background] Vermeulen A, Verdonck L, Kaufman JM. A critical evaluation of simple methods for the estimation of free testosterone in serum. J Clin Endocrinol Metab. 1999 Oct;84(10):3666-72. doi: 10.1210/jcem.84.10.6079. PMID 10523012
- [Background] Legro RS, Castracane VD, Kauffman RP. Detecting insulin resistance in polycystic ovary syndrome: purposes and pitfalls. Obstet Gynecol Surv. 2004 Feb;59(2):141-54. doi: 10.1097/01.OGX.0000109523.25076.E2. PMID 14752302